CLINICAL TRIAL: NCT06495502
Title: REVEAL To Disclose a Child Sexual Abuse Within Child & Adolescent Psychiatry Services: a Qualitative Study
Brief Title: To Disclose a Child Sexual Abuse Within Child & Adolescent Psychiatry Services
Acronym: REVEAL
Status: Recruiting | Type: Observational
Sponsor: Anne Revah-Levy (Other)
Responsible Party: Sponsor-Investigator, Anne Revah-Levy, Professor of child & adolescent psychiatry, Centre Hospitalier Victor Dupouy
Organization: Centre Hospitalier Victor Dupouy (Other)
Other Study IDs: CHVictorDupouy
Record Dates: First submitted 2024-06-27; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Child Sexual Abuse
Keywords: qualitative research; disclosure; child & adolescent psychiatry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients: i. be in a well-identified care path ii. Age: 12-25 years old iii. have experienced CSA iv. Child & adolescent psychiatry treatment prior to majority and after CSA, regardless the reason for this treatment v. No acute symptoms
  Interventions: Other: semi-structured interview
- Parents: i. child on a well-identified care path ii. child victim of CSA iii. Child disclosure during child & adolescent psychiatry treatment iv. not being the perpetrator in case of intrafamilial CSA perpetrated by the mother or the father (the other parent could be included).
  Interventions: Other: semi-structured interview
- child & adolescent mental health professionals: i. have experienced, directly or indirectly, at least one situation of CSA disclosure by a minor patient.
  Interventions: Other: semi-structured interview

INTERVENTIONS:
Other: semi-structured interview — Semi-structured interviews by qualitative health researchers

SUMMARY:
Mental health professionals investigating child sexual abuse (CSA) among children and adolescents is a major public health challenge. Many studies have shown the obstacles to disclose, with professionals having difficulties to address this issue and survivors having difficulties to disclose. Many children, old enough to tell what happened to them, would disclose this traumatic event only many years after, but they suffer from psychiatric and/or somatic disorders meanwhile. CSA survivors presenting psychiatric symptoms very often receive a psychiatric treatment within child & adolescent psychiatric (CAP) departments.

The investigators aim to better understand what is at stakes around the issue of disclosure of CSA by teenagers within CAP services, so to draw concrete implications to improve investigation efficacy and disclosure support by mental health professionals. To date, no study has ever explored these issues of investigating and disclosing CSA in CAP services. Qualitative methods are quite relevant here, aiming as they do, to in-depth explore complex issues, through the lived experience of the stakeholders.

The main objective of this study is to explore the lived experience of disclosing CSA among (i) adolescents and young adults followed in a CAP service, (ii) parents, and (iii) child & adolescent mental health professionals working in CAP services who have experienced a CSA disclosure. Crossing perspectives will bring answers to the complex question: "how to disclose a CSA within a CAP service?" and will lead to concrete implications to improve treatment of children and adolescents with an history of CSA.

It is an exploratory qualitative multi-center design following the IPSE approach - Inductive Process to analyze the structure of lived experience-.

DETAILED DESCRIPTION:
Mental health professionals investigating child sexual abuse (CSA) among children and adolescent is a major public health challenge. Many studies have shown the obstacles to disclose, with professionals having difficulties to address this issue and survivors having difficulties to disclose. Many children, old enough to tell what happened to them, would disclose this traumatic event only many years after, but they suffer from psychiatric and/or somatic disorders meanwhile. CSA survivors presenting psychiatric symptoms very often receive a psychiatric treatment within child & adolescent psychiatric (CAP) departments. This follow-up is to be considered as an opportunity for them to disclose. Yet, according to the current literature, 20% of women and 39% of men would not disclose the CSA. Among children and adolescents, disclosure rate is estimated between 16 and 25%. Reducing disclosure delay and improving the quality of mental health professionals support around the issue of disclosure and its outcomes (individual, family, forensic), could improve survivors prognostic.

The investigators aim to better understand what is at stakes around the issue of disclosure of CSA by teenagers within CAP services, so to draw concrete implications to improve investigation efficacy and disclosure support by mental health professionals. To date, no study ever explored these issues of investigating and disclosing CSA in CAP services. Qualitative methods are quite relevant here, aiming as they do, to in-depth explore complex issues, through the lived experience of the stakeholders.

The main objective of this study is to explore the lived experience of disclosing CSA among (i) adolescents and young adults followed in a CAP service, (ii) parents, and (iii) child & adolescent mental health professionals working in CAP services who have experienced a CSA disclosure. Crossing perspectives will bring answers to the complex question: "how to disclose a CSA within a CAP service?" and will lead to concrete implications to improve treatment of children and adolescents with an history of CSA.

It is an exploratory qualitative multi-center design following the IPSE approach - Inductive Process to analyze the structure of lived experience-. IPSE is a five-steps process: 1) set up a research group, 2) ensure the originality of the research, 3) organize recruitment and sampling intended to optimize exemplarity, 4) collect data that enable entry into the subjects 'experience, and 5) analyze the data. This final stage is composed of one individual descriptive phase, followed by two group phases: i) define the structure of the lived experience, and ii) translate the findings into concrete proposals that make a difference in care.

1 - Patients : i. be in a well-identified care path ii. Age: 12-25 years old iii. have experienced CSA iv. Child & adolescent psychiatry treatment prior to majority and after CSA, regardless the reason for this treatment v. No acute symptoms 2. Parents i. child on a well-identified care path ii. child victim of CSA iii. Child disclosure during child & adolescent psychiatry treatment iv. not being the perpetrator in case of intrafamilial CSA perpetrated by the mother or the father (the other parent could be included).

3. Child & adolescent mental health professionals i. have experienced, directly or indirectly, at least one situation of CSA disclosure by a minor patient.

This is a qualitative study, the number of participants required cannot be known beforehand, as it will be determined by the data saturation, based on the principle of theoretical sufficiency.

However, our experience in qualitative research allows us to propose a minimum of 30 participants per subgroup, for a total of 90 participants. This sample size will provide better visibility of our work and will ensure theoretical sufficiency.

Recruitment by local coordinators/co-investigators Data collection will be taken place within the five French departments.

The multicentric aspect is only to facilitate recruitment and to ensure data saturation but, in a qualitative study, it does not impact the quality and originality of the findings Intentional and non-probabilistic sampling strategy known as "Purposive Sampling" in maximum variation, that is to select exemplary/archetypal situations reflecting a variety of experiences, in order to obtain rich and diverse narratives, according to the principle of maximum variation. This is the technique of choice for sampling in qualitative research.

Data will be collected through semi-structured interviews by qualitative health researchers

All participants will be fully informed - orally and in writing- about the research and will express their non-opposition to participate in such research.

Non-opposition of the participants collected by the researcher and confirmed on the information and non-opposition form signed before any data collection and interview.

ELIGIBILITY:
Inclusion criteria:

* Adolescents and young adults from four child & adolescent psychiatric services in Argenteuil (SUPADO), Rouen, Lyon, Colombes and Rennes. T
* in a well-identified care path
* Age: 12-25 years old
* have experienced Child Sexual Abuse (CSA)
* Child & adolescent psychiatry treatment prior to majority and after CSA, regardless the reason for this treatment
* Parents with a Son/daughter on a well-identified care path, victim of CSA, with a disclosure during child & adolescent psychiatry treatment
* Child & adolescent mental health professionals

Exclusion criteria

* for adolescents, acute symptoms
* for parents, in the situation of intrafamily CSA perpetrated by a parent, this parent will be excluded

Ages: 12 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: The population under study is divided into three sub-groups
  * (1) adolescents and young adults aged between 12 and 25, CSA victims, who have been receiving child & adolescent psychiatry treatment.
  * (2) victim parents with an history of disclosure within the child & adolescent psychiatry treatment.
  * (3) Child & adolescent mental health professionals who have experienced, directly or indirectly, at least one situation of CSA disclosure by a minor patient.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Lived experience of disclosure of child sexual abuse | 2 years
  Participant-reported experiences in child sexual abuse disclosure as assessed using the Inductive Process to analyze the Structure of lived Experience (IPSE)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Sibeoni, MD PhD, Principal Investigator — Centre Hospitalier Victor Dupouy
Locations (5):
- France (5):
  - Hôpital Louis Mourier, Colombes, Hauts De Seine
  - Pôle Hospitalo-Universitaire de Psychiatrie de l'enfant et l'adolescent de Rennes, Rennes, Ille-et-Vilaine
  - Hopital Femme Mère Enfant, Hospices Civils de Lyon, Bron, Rhone
  - CHU Rouen/CH Rouvray, Rouen, Seine Maritime
  - CHVictorDupouy, Argenteuil, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No
anonymized data